CLINICAL TRIAL: NCT05453942
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Tolerability and Clinical Response After 4-week Oral Treatment With SAR441566 Compared With Placebo in Participants With Mild to Moderate Psoriasis
Brief Title: A Study to Investigate Safety, Tolerability and Clinical Response With SAR441566 Compared With Placebo in Participants With Mild to Moderate Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDY16918; U1111-1275-0915 (Registry Identifier: ICTRP); 2022-000850-27 (EudraCT Number)
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAR441566 (Experimental): Repeated dose of SAR441566 administered twice a day (BID) for 4 weeks under fed conditions
  Interventions: Drug: SAR441566
- Placebo (Placebo Comparator): Repeated dose of matching placebo administered twice a day (BID) for 4 weeks under fed condition
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR441566 — Repeated dose of SAR441566 administered twice a day (BID) for 4 weeks under fed conditions
  Arms: SAR441566
Drug: Placebo — Repeated dose of matching placebo administered twice a day (BID) for 4 weeks under fed condition
  Arms: Placebo

SUMMARY:
This is a parallel, Phase 1, single center, 2-arm, double-blind, randomized, placebo-controlled with a ratio 2 active: 1 placebo study for treatment of mild to moderate psoriasis participants. Approximately 36 participants (24 in the SAR441566 group and 12 in the placebo group) are to be enrolled to have a total of 33 evaluable participants (22 in the SAR441566 group and 11 in the placebo group).

The objective of this study is primarily to evaluate the tolerability and safety and secondarily the clinical response over 4-week oral treatment with SAR441566 in participants with mild to moderate psoriasis. The clinical response is measured by the relative change from baseline in Total Lesion Severity Score (TLSS).

The study comprises an up to 4-week screening period, a 4-week treatment period with SAR441566 or placebo. The end-of-study visit will be carried out 10 ±3 days after the last investigational medicinal product administration. The frequency of visits is once a week during the treatment period.

DETAILED DESCRIPTION:
* Screening period: up to 4 weeks
* Treatment: 4 weeks (from Day 1 to Day 28)
* End-of-Study: between 7 to 13 days after the last IMP administration (from Day 35 to Day 41) Total study duration: 37 to 69 days maximum (approximately between 6 and 10 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Male or female with mild to moderate psoriatic participants, between 18 and 65 years of age, inclusive.
* Body mass index between 18.0 and 35.0 kg/m2, inclusive (body weight not under 50.0 Kg).
* Female participants who are only postmenopausal or are sterilized (e.g post-bilateral surgical oophorectomy not linked to a history of cancer) can be included in the study.
* Participant must be in good health (except for psoriasis) as judged by the investigator, based on medical history, physical examination, vital signs, ECG, clinical laboratories, and urinalysis.
* Confirmed diagnosis of chronic plaque-type psoriasis, diagnosed at least 6 months prior to screening with mild to moderate severity, defined as PASI ≤ 16.
* Participant must have at least two lesions with TLSS≥4 at both screening and baseline excluding the scalp.

Exclusion Criteria:

* Pre-existing signs of skin atrophy, telangiectasia or striae in the affected area
* Use of systemic immunosuppressants within 4 weeks of entering the study and during the entire study duration
* Current evidence of non-plaque forms of psoriasis (e.g., erythrodermic, guttate or pustular), psoriatic arthritis
* Currently evidence or suspicion of drug-induced psoriasis (e.g., new onset or exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Use of any of the following therapies within 4 weeks prior to Baseline (Day 1): systemic non-biologic psoriasis therapies (including, but not limited to): psoralens and ultraviolet A (PUVA) therapy, cyclosporine, methotrexate, azathioprine, corticosteroids, apremilast, tofacitinib, oral retinoids, mycophenolate mofetil, sirolimus; or phototherapy (including UVB or self-treatment with tanning beds or therapeutic sunbathing) or topical psoriasis therapy with psoralens
* Use of topical corticosteroid preparations (except hydrocortisone 1%), topical calcineurin inhibitors, or other topical preparations with immunomodulatory properties within 2 weeks prior to randomization (Day 1)
* Prior use of any biologicals for treatment of psoriasis
* Participants who received any live vaccination within 3 months, any initial non-live vaccination within 30 days or non-live booster vaccination within 14 days of first IMP administration or intend to receive any vaccination during the study.
* Evidence of any clinically significant, severe or unstable, acute or chronically progressive, uncontrolled infection or medical condition (including an ongoing biological proven SARS-CoV-2 infection and recurrent infection) or any condition that may affect participant safety in the judgment of the Investigator including participants who are not adequately vaccinated against a SARS-CoV-2 infection according to local regulations.
* Opportunistic infections within 6 months before randomization (Day 1)

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAE) including SAE and AESI | Up to 69 days
  Assessment of adverse events (AE) / treatment-emergent adverse events (TEAE) including SAE and AESI

SECONDARY OUTCOMES:
Percent change from baseline in the target lesion severity score (TLSS) to weeks 2 and 4 | Baseline to week 4
  TLSS consists of a sum score of 3 clinical severity parameters (scaling, erythema, plaque elevation/induration; each graded on a 5-point severity scale; 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe/very severe) with a sum score ranging between 0 and 12 points

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number :2760001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PDY16918 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25321&tenant=MT_SNY_9011